CLINICAL TRIAL: NCT02928549
Title: Factors Associated With the Use of a High Volume Cancer Center by Black Women With Ovarian Cancer: A Qualitative Study
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1378
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: interviews; 16-1378
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Black Women with Cancer: In this formative qualitative research study we aim to use one-on-one semi-structured interviews with Black women diagnosed with ovarian cancer to learn about their experiences and their journey to accessing care at a high-volume ovarian cancer care center (HVC).
  Interventions: Behavioral: semi-structured interviews

INTERVENTIONS:
Behavioral: semi-structured interviews

SUMMARY:
The purpose of this study is to explore the experiences of Black women who receive care for ovarian cancer at Memorial Sloan Kettering Cancer Center, or "MSK" for short. The study consists of interviews with Black women who recently obtained some part of their ovarian cancer care at MSK.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have been diagnosed with ovarian, fallopian tube or primary peritoneal cancer and treated by an MSK physician.
* Participants must be able to provide verbal informed consent.
* Participants must be 18 years of age or older.
* Participants must self-identify as Black/African American.
* Participant must be able to understand and speak in English

Exclusion Criteria:

* Inability or refusal to identify race/ethnicity.
* Presence or development of a physical, cognitive or psychiatric deficit resulting in an inability to provide meaningful informed consent or to understand the study or complete the interview.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK Gynecology clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
accessing care | 1 year
  The study team will review and code the interview transcripts through a process of independent and collaborative thematic content analysis,[15-18] using ATLAS.ti (a qualitative data analysis software package) to facilitate the analysis process.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Long-Roche, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/